CLINICAL TRIAL: NCT01321567
Title: Quality of Life in New Treatable Therapy as Rabeprazole Option for Refractory Reflux Esophagitis
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: PRT11T
Record Dates: First submitted 2011-03-18; First posted 2011-03-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2015-05

CONDITIONS: Refractory Reflux Esophagitis
Keywords: rabeprazole sodium; refractory reflux esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rabeprazole Sodium
  Interventions: Drug: rabeprazole sodium

INTERVENTIONS:
Drug: rabeprazole sodium — Doses of 10 mg or 20 mg twice daily may be administered orally to reflux esophagitis patients for a further 8 weeks when proton pump inhibitor treatment is ineffective. However, a dose of 20 mg twice daily should only be administered to patients with severe mucosa injury.

SUMMARY:
To investigate the efficacy and safety of PARIET twice daily (b.i.d.) in patients with Proton Pump Inhibitor-resistant reflux esophagitis

ELIGIBILITY:
Inclusion criteria;

-Proton pump inhibitor-resistant reflux esophagitis. (Patients who have mucosal breaks (erosions, ulcers) on endoscopy)

Exclusion criteria;

* Patients with a history of hypersensitivity to any ingredients of PARIET.
* Patients on atazanavir sulfate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals and Clinics in Japan
Sampling Method: Non-Probability Sample
Enrollment: 2157 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with improvement based on health related Quality of Life (QOL) questionnaire | Check at predose, 4, 8, 16 and 32 weeks

SECONDARY OUTCOMES:
Number of subjects with improvement in symptoms of GERD | Check at predose, 4, 8, 16 and 32 weeks
Endoscopic healing rate | 8 weeks
Adverse events | Every 4-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshinori Furuhata, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Regulatory Compliance, Safety and Quality Assurance Headquarters, Eisai Co., Ltd.
Locations (447):
- Japan (447):
  - Aisai, Aichi-ken
  - Anjo, Aichi-ken
  - Gamagōri, Aichi-ken
  - Ichinomiya, Aichi-ken
  - Inuyama, Aichi-ken
  - Kariya, Aichi-ken
  - Kasugai, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Owariasahi, Aichi-ken
  - Tokoname, Aichi-ken
  - Toyota, Aichi-ken
  - Tōkai, Aichi-ken
  - Tsushima, Aichi-ken
  - Daisen, Akita
  - Yokote, Akita
  - Yurihonjō, Akita
  - Goshogawara, Aomori
  - Hachinohe, Aomori
  - Hirosaki, Aomori
  - Kitatsugaru, Aomori
  - Mutsu, Aomori
  - Sannohe, Aomori
  - Towada, Aomori
  - Asahi, Chiba
  - Choshi, Chiba
  - Funabashi, Chiba
  - Ichihara, Chiba
  - Ichikawa, Chiba
  - Kashiwa, Chiba
  - Katori-shi, Chiba
  - Matsudo, Chiba
  - Mobara, Chiba
  - Narashino, Chiba
  - Noda, Chiba
  - Imabari, Ehime
  - Kitauwa, Ehime
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Ōzu, Ehime
  - Saijō, Ehime
  - Uwajima, Ehime
  - Mikatakaminaka, Fukui
  - Ono, Fukui
  - Sabae, Fukui
  - Sakai, Fukui
  - Asakura, Fukuoka
  - Buzen, Fukuoka
  - Chikushi, Fukuoka
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Miyama, Fukuoka
  - Munakata, Fukuoka
  - Nōgata, Fukuoka
  - Omuta, Fukuoka
  - Ōkawa, Fukuoka
  - Tagawa, Fukuoka
  - Tsuiki, Fukuoka
  - Wakasugi, Fukuoka
  - Yame, Fukuoka
  - Iwaki, Fukushima
  - Kōriyama, Fukushima
  - Shirakawa, Fukushima
  - Sōma, Fukushima
  - Yama, Fukushima
  - Hashima, Gifu
  - Kakamigahara, Gifu
  - Minokamo, Gifu
  - Mizunami, Gifu
  - Ōgaki, Gifu
  - Sekimachi, Gifu
  - Tajimi, Gifu
  - Takayama, Gifu
  - Agatsuma, Gunma
  - Kiryū, Gunma
  - Maebashi, Gunma
  - Midori, Gunma
  - Ōta, Gunma
  - Takasaki, Gunma
  - Aki, Hiroshima
  - Fukuyama, Hiroshima
  - Higashihiroshima, Hiroshima
  - Kure, Hiroshima
  - Mihara, Hiroshima
  - Miyoshi, Hiroshima
  - Onomichi, Hiroshima
  - Takehara, Hiroshima
  - Abashiri, Hokkaido
  - Abuta, Hokkaido
  - Asahikawa, Hokkaido
  - Date, Hokkaido
  - Ebetsu, Hokkaido
  - Eniwa, Hokkaido
  - Fukagawa, Hokkaido
  - Furano, Hokkaido
  - Hakodate, Hokkaido
  - Hokuto, Hokkaido
  - Ishikari, Hokkaido
  - Kamiiso, Hokkaido
  - Kasai, Hokkaido
  - Kato, Hokkaido
  - Kayabe, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Muroran, Hokkaido
  - Nakagawa, Hokkaido
  - Obihiro, Hokkaido
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Shibetsu, Hokkaido
  - Suttsu, Hokkaido
  - Tomakomai, Hokkaido
  - Yoichi, Hokkaido
  - Aioi, Hyōgo
  - Akashi, Hyōgo
  - Ako, Hyōgo
  - Amagasaki, Hyōgo
  - Ashiya, Hyōgo
  - Awaji, Hyōgo
  - Himeji, Hyōgo
  - Itami, Hyōgo
  - Kakogawa, Hyōgo
  - Kobe, Hyōgo
  - Miki, Hyōgo
  - Nishinomiya, Hyōgo
  - Ono, Hyōgo
  - Sanda, Hyōgo
  - Sasayama, Hyōgo
  - Sumoto, Hyōgo
  - Takarazuka, Hyōgo
  - Tamba, Hyōgo
  - Bandō, Ibaraki
  - Hitachi, Ibaraki
  - Hitachiota, Ibaraki
  - Hokota, Ibaraki
  - Ishioka, Ibaraki
  - Itako, Ibaraki
  - Jōsō, Ibaraki
  - Kitaibaraki, Ibaraki
  - Koga, Ibaraki
  - Mito, Ibaraki
  - Moriya, Ibaraki
  - Naka, Ibaraki
  - Ryūgasaki, Ibaraki
  - Shimo-tsuma, Ibaraki
  - Tsukuba, Ibaraki
  - Ushiku, Ibaraki
  - Hakui, Ishikawa-ken
  - Hakusan, Ishikawa-ken
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Nomi, Ishikawa-ken
  - Hanamaki, Iwate
  - Ichinoseki, Iwate
  - Morioka, Iwate
  - Ōshū, Iwate
  - Tōno, Iwate
  - Kan’onjichō, Kagawa-ken
  - Marugame, Kagawa-ken
  - Mitoyo, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Aira, Kagoshima-ken
  - Ichikikushikino, Kagoshima-ken
  - Isa, Kagoshima-ken
  - Izumi, Kagoshima-ken
  - Kanoya, Kagoshima-ken
  - Kirishima, Kagoshima-ken
  - Kumage, Kagoshima-ken
  - Sendai, Kagoshima-ken
  - Ashigarashimo, Kanagawa
  - Atsugi, Kanagawa
  - Chigasaki, Kanagawa
  - Fujisawa, Kanagawa
  - Hadano, Kanagawa
  - Hiratsuka, Kanagawa
  - Isehara, Kanagawa
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Minamiashigara, Kanagawa
  - Naka, Kanagawa
  - Odawara, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Zama, Kanagawa
  - Aso, Kumamoto
  - Hitoyoshi, Kumamoto
  - Isshōchi, Kumamoto
  - Kamimashiki, Kumamoto
  - Kōshi, Kumamoto
  - Yatsushiro, Kumamoto
  - Fukuchiyama, Kyoto
  - Kameoka, Kyoto
  - Kyōtango, Kyoto
  - Maizuru, Kyoto
  - Mukō, Kyoto
  - Nantan, Kyoto
  - Yosa, Kyoto
  - Iga, Mie-ken
  - Ise, Mie-ken
  - Kameyama, Mie-ken
  - Kitamuro, Mie-ken
  - Kuwana, Mie-ken
  - Matsusaka, Mie-ken
  - Suzuka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Shiroishi, Miyagi
  - Toda, Miyagi
  - Tome, Miyagi
  - Ebino, Miyazaki
  - Hyūga, Miyazaki
  - Koyu, Miyazaki
  - Kushima, Miyazaki
  - Miyakonojō, Miyazaki
  - Nobeoka, Miyazaki
  - Ina, Nagano
  - Kamiina, Nagano
  - Kiso, Nagano
  - Komagane, Nagano
  - Matsumoto, Nagano
  - Nakano, Nagano
  - Saku, Nagano
  - Ueda, Nagano
  - Isahaya, Nagasaki
  - Sasebo, Nagasaki
  - Unzen, Nagasaki
  - Gojō, Nara
  - Ikoma, Nara
  - Kashihara, Nara
  - Kitakatsuragi, Nara
  - Ōuda-yamaguchi, Nara
  - Sakurai, Nara
  - Tenri, Nara
  - Yamatokōriyama, Nara
  - Yamatotakada, Nara
  - Jōetsu, Niigata
  - Kashiwazaki, Niigata
  - Minamiuonuma, Niigata
  - Mitsuke, Niigata
  - Nagaoka, Niigata
  - Sado, Niigata
  - Shibata, Niigata
  - Tōkamachi, Niigata
  - Kunisaki, Oita Prefecture
  - Nakatsu, Oita Prefecture
  - Taketa, Oita Prefecture
  - Usa, Oita Prefecture
  - Yufu, Oita Prefecture
  - Akaiwa, Okayama-ken
  - Asakuchi, Okayama-ken
  - Bizen, Okayama-ken
  - Kurashiki, Okayama-ken
  - Niimi, Okayama-ken
  - Tsukubo, Okayama-ken
  - Tsuyama, Okayama-ken
  - Itoman, Okinawa
  - Nago, Okinawa
  - Nakagami, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Daitō, Osaka
  - Fujiidera, Osaka
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Ibaraki, Osaka
  - Izumi, Osaka
  - Izumiōtsu, Osaka
  - Izumisano, Osaka
  - Kadoma, Osaka
  - Katano, Osaka
  - Kishiwada, Osaka
  - Matsubara, Osaka
  - Minamikawachi, Osaka
  - Mino, Osaka
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Sennan, Osaka
  - Settsu, Osaka
  - Suita, Osaka
  - Takaishi, Osaka
  - Takatsuki, Osaka
  - Tondabayashi, Osaka
  - Toyonaka, Osaka
  - Yao, Osaka
  - Imari, Saga-ken
  - Kanzaki, Saga-ken
  - Ogi, Saga-ken
  - Takeo, Saga-ken
  - Taku, Saga-ken
  - Tosu, Saga-ken
  - Ageo, Saitama
  - Chichibu, Saitama
  - Fujimi, Saitama
  - Fukaya, Saitama
  - Hannō, Saitama
  - Hidaka, Saitama
  - Kasukabe, Saitama
  - Kawagoe, Saitama
  - Kawaguchi, Saitama
  - Kazo, Saitama
  - Kitaadachi, Saitama
  - Koshigaya, Saitama
  - Kukichūō, Saitama
  - Sayama, Saitama
  - Toda, Saitama
  - Tokorozawa, Saitama
  - Warabi, Saitama
  - Kōka, Shiga
  - Kusatsu, Shiga
  - Moriyama, Shiga
  - Nagahama, Shiga
  - Ōtsu, Shiga
  - Rittō, Shiga
  - Izumo, Shimane
  - Matsue, Shimane
  - Yasugi, Shimane
  - Fuji, Shizuoka
  - Fujieda, Shizuoka
  - Fujinomiya, Shizuoka
  - Fukuroi, Shizuoka
  - Hamamatsu, Shizuoka
  - Itō, Shizuoka
  - Iwata, Shizuoka
  - Kikugawa, Shizuoka
  - Mishima, Shizuoka
  - Numazu, Shizuoka
  - Shimada, Shizuoka
  - Shimoda, Shizuoka
  - Susono, Shizuoka
  - Yaizu, Shizuoka
  - Mooka, Tochigi
  - Nikkō, Tochigi
  - Sano, Tochigi
  - Shimotsuga, Tochigi
  - Utsunomiya, Tochigi
  - Anan, Tokushima
  - Awa, Tokushima
  - Myozai, Tokushima
  - Narutochō-mitsuishi, Tokushima
  - Okuno, Tokushima
  - Adachi City, Tokyo
  - Akiruno, Tokyo
  - Akishima, Tokyo
  - Bunkyo, Tokyo
  - Chiyoda City, Tokyo
  - Chūō, Tokyo
  - Edogawa City, Tokyo
  - Fuchū, Tokyo
  - Hachiōji, Tokyo
  - Higashimurayama, Tokyo
  - Higashiyamato, Tokyo
  - Hino, Tokyo
  - Inagi, Tokyo
  - Katsushika-ku, Tokyo
  - Kita-ku, Tokyo
  - Kodaira, Tokyo
  - Koganei, Tokyo
  - Koto, Tokyo
  - Machida, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Mitaka, Tokyo
  - Nakano City, Tokyo
  - Nerima City, Tokyo
  - Nishitōkyō, Tokyo
  - Ōme, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - Suginami, Tokyo
  - Sumida City, Tokyo
  - tabashi City, Tokyo
  - Tachikawa, Tokyo
  - Toshima City, Tokyo
  - Kurayoshi, Tottori
  - Sakaiminato, Tottori
  - Imizu, Toyama
  - Kurobe-shi, Toyama
  - Nakaniikawa, Toyama
  - Namerikawa, Toyama
  - Nanto, Toyama
  - Takaoka, Toyama
  - Tonami, Toyama
  - Gobō, Wakayama
  - Higashimuro, Wakayama
  - Iwade, Wakayama
  - Kainan, Wakayama
  - Nishimuro, Wakayama
  - Tanabe, Wakayama
  - Higashiokitama, Yamagata
  - Kaminoyama, Yamagata
  - Sakata, Yamagata
  - Hagi, Yamaguchi
  - Hikari, Yamaguchi
  - Iwakuni, Yamaguchi
  - Sanyōonoda, Yamaguchi
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi
  - Yanai, Yamaguchi
  - Chūō, Yamanashi
  - Fuefuki, Yamanashi
  - Kofu, Yamanashi
  - Kōshū, Yamanashi
  - Minami-Alps, Yamanashi
  - Minamikoma, Yamanashi
  - Tsuru, Yamanashi
  - Aichi
  - Akita
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Mie
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nara
  - Niigata
  - Okayama
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokushima
  - Tottori
  - Toyama
  - Wakayama
  - Yamagata
  - Yamanashi

REFERENCES:
- [Result] Kinoshita Y, Hongo M, Kusano M, Furuhata Y, Miyagishi H, Ikeuchi S; RPZ Study Group. Therapeutic Response to Twice-daily Rabeprazole on Health-related Quality of Life and Symptoms in Patients with Refractory Reflux Esophagitis: A Multicenter Observational Study. Intern Med. 2017;56(10):1131-1139. doi: 10.2169/internalmedicine.56.7896. Epub 2017 May 15. PMID 28502925